CLINICAL TRIAL: NCT01146158
Title: Individualisation of the Lymphatic Arm Drainage During Axillary Dissection for Breast Carcinomas.
Brief Title: Axillary Reverse Mapping for Breast Carcinomas
Acronym: SENTIBRAS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P070154
Record Dates: First submitted 2010-04-23; First posted 2010-06-17 (Estimated); Last update posted 2015-04-08 (Estimated); Status verified 2009-05

CONDITIONS: Axillary Dissection
Keywords: Axillary dissection

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- surgery Axillary dissection (Experimental): surgery Axillary dissection
  Interventions: Procedure: Axillary dissection for breast carcinomas

INTERVENTIONS:
Procedure: Axillary dissection for breast carcinomas — surgery Axillary dissection
  Other Names: surgery Axillary dissection

SUMMARY:
Distinct arm from breast axillary dissection (AD), or axillary reverse mapping (ARM), involves retrieving all breast related nodes while leaving intact the main lymphatic drainage chain of the upper limb. This represents a new surgical technique that is the focus of recent surgical interest.

DETAILED DESCRIPTION:
Distinct arm from breast axillary dissection (AD), or axillary reverse mapping (ARM), involves retrieving all breast related nodes while leaving intact the main lymphatic drainage chain of the upper limb. This represents a new surgical technique that is the focus of recent surgical interest. The assumption is that the sentinel node (SN) of the upper limb is different from the SN of the breast and that it is uninvolved after metastatic involvement of the axillary nodes in relation to the breast. During the ARM procedure, it is necessary to use an injection of a lymphatic tracer into the upper limb in order to visualize the lymphatic arm drainage.The ultimate goal for ARM procedure is to reduce the rate of lymphedema in N+ patients requiring an AD.

ELIGIBILITY:
Inclusion Criteria:

* Indication for formal Axillary Dissection (AD)
* N0 patient with a large tumor: T3
* N1 patient
* N2 patient with axillary imaging showing limited node involvement(1-4N+).
* Secondary AD after a positive sentinel node ( pN1, pN1(mi))
* AD after préopérative chemotherapy in a patient initially N+.
* Age between 18 and 70
* Signature of the consent form.
* Patients beneficiary of the Social Security

Exclusion Criteria:

* N0 patient with an indication of Sentinel Node biopsy
* N2 patient with axillary imaging showing suspected node involvement >4N+.
* N3 patient
* Age over 70
* Pregnancy
* Blue dye allergy
* Mentally deficient patient

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Actual)
Dates: Start 2009-11; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Success of the principal objectives is qualified as finding one or more radioactive node in zone D | 1 day
  Zone D is the area lateral to the lateral thoracic vein and extending from the second intercostobrachial nerve to the axillary vein.
  If all radioactive nodes are found below the second intercostobrachial nerve (Zone C, A) or medial to the lateral thoracic vein (Zone A, B) this qualifies a failure of the main objective

SECONDARY OUTCOMES:
Evaluate the incidence of metastatic or micro-metastatic disease within the "SENTIBRAS " node | 15 days
  Evaluate the incidence of metastatic or micro-metastatic disease within
Evaluate the correlation between clinical and histological results | 15 days
  Evaluate the correlation between clinical and histological results
Evaluate the morbidity associated with Axillary Dissection. | 1 year, 2 years and 5 years
  Evaluate the morbidity associated with Axillary Dissection.

CONTACTS AND LOCATIONS:
Overall Officials: Claude NOS, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hospital European Georges Pompidou, Paris, France

REFERENCES:
- [Background] Nos C, Lesieur B, Clough KB, Lecuru F. Blue dye injection in the arm in order to conserve the lymphatic drainage of the arm in breast cancer patients requiring an axillary dissection. Ann Surg Oncol. 2007 Sep;14(9):2490-6. doi: 10.1245/s10434-007-9450-4. Epub 2007 Jun 5. PMID 17549570
- [Background] Nos C, Kaufmann G, Clough KB, Collignon MA, Zerbib E, Cusumano P, Lecuru F. Combined axillary reverse mapping (ARM) technique for breast cancer patients requiring axillary dissection. Ann Surg Oncol. 2008 Sep;15(9):2550-5. doi: 10.1245/s10434-008-0030-z. Epub 2008 Jul 11. PMID 18618185